CLINICAL TRIAL: NCT01880320
Title: A Multi-center, Randomized, Double-blind, Parallel-group Vehicle and Active Controlled Study to Compare the Efficacy and Safety of CD0271 0.3% / CD1579 2.5% Topical Gel Versus Topical Gel Vehicle in Subjects With Acne Vulgaris
Brief Title: Multi-center, Randomized, Double-blind Efficacy and Safety of CD0271 0.3%/CD1579 2.5 % Topical Gel in Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.06.SPR.18240
Record Dates: First submitted 2013-06-14; First posted 2013-06-18 (Estimated); Results first posted 2016-09-09 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CD0271 0.3% /CD1579 2.5% Gel (Experimental): active arm
  Interventions: Drug: CD0271 0.3% / CD1579 2.5%
- CD0271 0.1% / CD1579 2.5% (Active Comparator): Comparator arm
  Interventions: Drug: CD0271 0.1% / CD1579 2.5%
- Topical Gel Vehicle (Placebo Comparator): Placebo arm
  Interventions: Drug: Topical Gel Vehicle

INTERVENTIONS:
Drug: CD0271 0.3% / CD1579 2.5%
  Arms: CD0271 0.3% /CD1579 2.5% Gel
Drug: CD0271 0.1% / CD1579 2.5%
  Arms: CD0271 0.1% / CD1579 2.5%
Drug: Topical Gel Vehicle
  Arms: Topical Gel Vehicle

SUMMARY:
The study hypothesis are based on the assumption that :

* CD0271 0.3%/CD1579 2.5% Gel provides superior clinical efficacy compared with Topical Gel Vehicle in the overall population and in the subgroup of severe Subjects
* CD0271 0.3%/CD1579 2.5% Gel applied once daily for up to 12 weeks has an acceptable safety and tolerability profile

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, who is 12 years of age or older at Screening visit.
2. Clinical diagnosis of acne vulgaris with facial involvement.
3. An IGA of Moderate (3) or Severe (4) at Baseline visit.
4. A minimum of 20 but not more than 100 inflammatory lesions (papules and pustules) on the face (including the nose) at Baseline visit.
5. A minimum of 30 but not more than 150 non-inflammatory lesions (open comedones and closed comedones) on the face (including the nose) at Baseline visit.

Exclusion Criteria:

1. More than 2 acne nodules on the face at Baseline visit.
2. Acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.), nodulo cystic acne, or acne requiring systemic treatment.
3. Underlying diseases or other dermatologic conditions that require the use of interfering topical or systemic therapy or that might interfere with study assessments such as, but not limited to, atopic dermatitis, perioral dermatitis or rosacea. This includes clinically significant abnormal findings, uncontrolled or serious disease, or any medical or surgical condition, that may either interfere with the interpretation of the clinical trial results, and/or put the subject at significant risk (according to Investigator's judgment) if he/she participates in the clinical trial.
4. The subject has received, applied or taken some specified treatments within the specified timeframe prior to the Baseline visit
5. The subject is unwilling to refrain from use of prohibited medication during the clinical trial.
6. Use of hormonal contraceptives solely for control of acne.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (25):
  - Galderma Investigational site, Birmingham, Alabama
  - Galderma Investigationnal Site, Mobile, Alabama
  - Galderma investigational Site, Hot Springs, Arkansas
  - Galderma Investigational Site, Los Angeles, California
  - Galderma Investigational Site, Sacramento, California
  - Galderma Investigational Site, Santa Monica, California
  - Galderma Investigational Site, Miami, Florida
  - Galderma Investigational Site, Miramar, Florida
  - Galderma Investiogational Site, Newnan, Georgia
  - Galderma Investigational Site, Snellville, Georgia
  - Galderma Investigational Site, Chicago, Illinois
  - Galderma Investigational Site, Detroit, Michigan
  - Galderma Investigational Site, Albuquerque, New Mexico
  - Galderma Investigational Site, New York, New York
  - Galderma Investigational Site, Stony Brook, New York
  - Galderma Investigational Site, Raleigh, North Carolina
  - Galderma Investigational Site, Beachwood, Ohio
  - Galderma investigational Site, Hershey, Pennsylvania
  - Galderma Investigational Site, Greenville, South Carolina
  - Galderma Investigational Site, Goodlettsville, Tennessee
  - Galderma Investigational Site, Knoxville, Tennessee
  - Galderma Investigational Site, Arlington, Texas
  - Galderma Investigational Site, San Antonio, Texas
  - Galderma Investigational Site, Salt Lake City, Utah
  - Galderma Investigational Site, Spokane, Washington
- Canada (6):
  - Galderma Investigational Site, Barrie
  - Galderma Investigational Site, Markham
  - Galderma Investiogational Site, Montreal
  - Galderma Investigational Site, Peterborough
  - Galderma Investigational site, Surrey
  - Galderma Investigational Site, Waterloo

REFERENCES:
- [Derived] Stein Gold L, Werschler WP, Mohawk J. Adapalene/Benzoyl Peroxide Gel 0.3%/2.5%: Effective Acne Therapy Regardless of Age or Gender. J Drugs Dermatol. 2017 Jun 1;16(6):582-589. PMID 28686776
- [Derived] Alexis AF, Cook-Bolden FE, York JP. Adapalene/Benzoyl Peroxide Gel 0.3%/2.5%: A Safe and Effective Acne Therapy in All Skin Phototypes. J Drugs Dermatol. 2017 Jun 1;16(6):574-581. PMID 28686775
- [Derived] Stein Gold L, Weiss J, Rueda MJ, Liu H, Tanghetti E. Moderate and Severe Inflammatory Acne Vulgaris Effectively Treated with Single-Agent Therapy by a New Fixed-Dose Combination Adapalene 0.3 %/Benzoyl Peroxide 2.5 % Gel: A Randomized, Double-Blind, Parallel-Group, Controlled Study. Am J Clin Dermatol. 2016 Jun;17(3):293-303. doi: 10.1007/s40257-016-0178-4. PMID 26945741

RESULTS

PARTICIPANT FLOW:
Groups:
- CD0271 0.3% /CD1579 2.5% Gel: Active arm
  CD0271 0.3% / CD1579 2.5%
- CD0271 0.1% / CD1579 2.5%: Comparator arm
  CD0271 0.1% / CD1579 2.5%
- Topical Gel Vehicle: Placebo arm
  Topical Gel Vehicle
Period: Overall Study
Arm/Group | CD0271 0.3% /CD1579 2.5% Gel | CD0271 0.1% / CD1579 2.5% | Topical Gel Vehicle
Started | 217 | 217 | 69
Completed | 197 | 192 | 61
Not Completed | 20 | 25 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD0271 0.3% /CD1579 2.5% Gel | CD0271 0.1% / CD1579 2.5% | Topical Gel Vehicle | Total
Number analyzed (Participants) | 217 | 217 | 69 | 503
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 124 | 136 | 43 | 303
  Between 18 and 65 years | 93 | 81 | 26 | 200
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.1 (7.59) | 19.4 (6.75) | 18.5 (5.72) | 19.6 (7.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 114 | 36 | 263
  Male | 104 | 103 | 33 | 240
Region of Enrollment [Number; unit: participants]
  Canada | 17 | 16 | 5 | 38
  United States | 200 | 201 | 64 | 465
Baseline Investigator Global Assessment (IGA) [Number; unit: participants]
  Baseline IGA = Moderate (3) | 111 | 105 | 35 | 251
  Baseline IGA = Severe (4) | 106 | 112 | 34 | 252

OUTCOME MEASURES:

1. Primary Outcome: Success Rate
Description: Success was defined as 'Clear' or 'Almost Clear' on the Investigator Global Assessment (IGA).
  Success rate at Week 12 was estimated using multiple imputation approach which is an average of response from multiple imputed datasets.
Time Frame: Week 12
Population: Intent-to-treat (ITT): All subjects who were randomized. Baseline IGA Severe population: All randomized subjects who had IGA=4 at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | CD0271 0.3% /CD1579 2.5% Gel | CD0271 0.1% / CD1579 2.5% | Topical Gel Vehicle
Number analyzed (Participants) | 217 | 217 | 69
percentage of participants
  All subjects (MI: Multiple Imputation) | 33.7 | 27.3 | 11.0
  Baseline IGA=Severe (4) (MI: Multiple Imputation): number analyzed (Participants) | 106 | 112 | 34
  Baseline IGA=Severe (4) (MI: Multiple Imputation) | 31.9 | 20.5 | 11.8

2. Primary Outcome: Changes From Baseline in Inflammatory Lesion Counts
Time Frame: Baseline - Week12
Population: ITT Population, Multiple imputation
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | CD0271 0.3% /CD1579 2.5% Gel | CD0271 0.1% / CD1579 2.5% | Topical Gel Vehicle
Number analyzed (Participants) | 217 | 217 | 69
Lesions
  All Subjects | -27.04 (0.846) | -26.72 (0.822) | -14.40 (1.460)
  Baseline IGA = Severe (4): number analyzed (Participants) | 106 | 112 | 34
  Baseline IGA = Severe (4) | -35.17 (1.407) | -31.92 (1.320) | -15.46 (2.297)

3. Primary Outcome: Changes From Baseline in Non-Inflammatory Lesion Counts
Time Frame: Baseline - Week 12
Population: ITT Population, Multiple Imputation
Measure: Least Squares Mean (Standard Error); unit: lesions
Arm/Group | CD0271 0.3% /CD1579 2.5% Gel | CD0271 0.1% / CD1579 2.5% | Topical Gel Vehicle
Number analyzed (Participants) | 217 | 217 | 69
lesions
  All Subjects | -40.18 (1.332) | -39.00 (1.277) | -18.47 (2.270)
  Baseline IGA = Severe (4): number analyzed (Participants) | 106 | 112 | 34
  Baseline IGA = Severe (4) | -45.61 (2.058) | -43.10 (1.847) | -17.25 (3.337)

ADVERSE EVENTS:
Arm/Group | CD0271 0.3% /CD1579 2.5% Gel | CD0271 0.1% / CD1579 2.5% | Topical Gel Vehicle
Serious Adverse Events (participants affected / at risk) | 0/217 | 1/217 | 0/69
Other Adverse Events (participants affected / at risk) | 34/217 | 23/217 | 13/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD0271 0.3% /CD1579 2.5% Gel (N=217) | CD0271 0.1% / CD1579 2.5% (N=217) | Topical Gel Vehicle (N=69)
Generalized Anxiety Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CD0271 0.3% /CD1579 2.5% Gel (N=217) | CD0271 0.1% / CD1579 2.5% (N=217) | Topical Gel Vehicle (N=69)
Nasopharyngitis (Infections and infestations) | 14 | 11 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 5 | 4
Infleunza (Infections and infestations) | 2 | 2 | 1
Gastroenteritis (Infections and infestations) | 3 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 9 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Rhinitis seasonal (Nervous system disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No